CLINICAL TRIAL: NCT04466228
Title: Effects of Non-invasive Transcranial Electrical Stimulation on Cognition in Patients With Multiple Sclerosis
Brief Title: Non-invasive Transcranial Electrical Stimulation in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-1908-34831
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Stim1 high dose (Experimental): This group will receive high dose non-invasive transcranial electrical stimulation
  Interventions: Device: non-invasive transcranial electrical stimulation
- Stim2 low dose (Experimental): This group will receive low dose non-invasive transcranial electrical stimulation
  Interventions: Device: non-invasive transcranial electrical stimulation
- Sham control (Sham Comparator): This group will receive sham control non-invasive transcranial electrical stimulation
  Interventions: Device: non-invasive transcranial electrical stimulation

INTERVENTIONS:
Device: non-invasive transcranial electrical stimulation — Non-invasive transcranial electrical stimulation across the prefrontal cortex.

SUMMARY:
The goal is to investigate the effects of non-invasive transcranial electrical stimulation on cognition in MS.

DETAILED DESCRIPTION:
The participants' baseline cognitive function will be assessed with a tablet-based, videogame-like software specifically designed as a medical device to test and train cognitive function for populations with cognitive disorders. After baseline test assessment, participants will receive stimulation while playing the training version of the software. After the stimulation, cognitive performance will be evaluated again with the testing version. Investigators will assess changes in cognitive performance associated with stimulation.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65,
* diagnosis of MS
* Expanded Disability Status Scale (EDSS)≤6.5, no paresis of the upper limbs
* a minimum of 3 months since the last relapse
* Beck Depression Inventory<19
* normal hearing
* and no changes in MS or symptomatic medications in past 2 months

Exclusion Criteria:

* prior brain surgery
* clips in brain
* epilepsy or other neurological or non-affective psychiatric disorders
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Sandler Neurosciences Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu WY, Zanto T, Park JE, Gazzaley A, Bove RM. Effects of transcranial alternating current stimulation on cognitive function in people with multiple sclerosis: A randomized controlled trial. Mult Scler Relat Disord. 2023 Dec;80:105090. doi: 10.1016/j.msard.2023.105090. Epub 2023 Oct 19. PMID 37925960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stim1 High Dose | Stim2 Low Dose | Sham Control
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stim1 High Dose | Stim2 Low Dose | Sham Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (7.6) | 42.8 (9.3) | 47.4 (8.0) | 46.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 17 | 48
  Male | 3 | 6 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 14 | 11 | 15 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 3 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Processing Speed Change From Baseline Assessment
Description: Symbol Digit Modalities Test (SDMT) score will be used to measure processing speed. SDMT measures the time to pair abstract symbols with specific numbers. The test requires visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items in 90 seconds. (max=110, min=0). Higher scores indicate improvement. Lower scores indicate worsening.
Time Frame: Baseline (pre-stim) and post-stimulation (up to 2 hours)
Population: The present report covers all collected data. In a formal data analysis, three participants were excluded from the analyses: 2 due to poor performance at baseline (lower than 2 standard deviation of all 60 participants); and 1 for not following instructions properly during post-stim assessment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stim2 Low Dose | Stim1 High Dose | Sham Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale
  pre-stim | 41.65 (2.65) | 42.05 (2.68) | 44.4 (1.8)
  post-stim | 46.1 (2.81) | 44.8 (2.82) | 44.8 (1.4)

2. Primary Outcome: EVO Performance Change From Baseline Assessment
Description: EVO tool is a digital cognitive assessment developed to assess cognitive function including attention and related cognitive control processes in clinical populations. It comes with the closed-loop adaptive algorithm which makes proportional changes in gameplay difficulty when the participant's performance deviates from an 80% rate of accuracy, which ensures that task difficulty is equated across participants and enhances engagement. Gameplay threshold (level 0 to level 20), response time and response time variability will be measured to evaluate attention control. Higher threshold level, lower response time and smaller response time variability indicate improvement.
Time Frame: Baseline (pre-stim) and post-stimulation, up to 2 hours
Population: EVO performance change from baseline assessment was not measured in the study. Therefore the analysis was not performed.
Arm/Group | Stim1 High Dose | Stim2 Low Dose | Sham Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: At the end of the study session (10 minutes after the cessation of the stimulation).
Description: At the end of the study (10 minutes after the cessation of the stimulation)., all participants were asked to complete a survey rating their perception of stimulation (headache, neck pain, scalp pain, tingling, itching, burning sensation, sleepiness, trouble concentrating, and acute mood change, phosphene) on a Likert scale from 0 (none) to 10 (not tolerable).
Arm/Group | Stim1 High Dose | Stim2 Low Dose | Sham Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT04466228/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT04466228/ICF_001.pdf